CLINICAL TRIAL: NCT02199288
Title: A NON-INTERVENTIONAL STUDY TO EVALUATE THE EFFECTIVENESS, SAFETY AND NURSE MANAGEMENT DURING INDUCTION TREATMENT WITH MABTHERA S.C. FOLLOWING A FIRST INITIAL MABTHERA I.V. TREATMENT, IN PATIENTS WITH NON-HODGKINS LYMPHOMA IN A REAL-LIFE SETTING
Brief Title: Effectiveness, Safety & Nurse Management Study of MabThera SC in Patients With Non-Hodgkin's Lymphoma: Real-Life Setting
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29314
Record Dates: First submitted 2014-07-18; First posted 2014-07-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective, open-label, multicenter, observational study will investigate the effectiveness and safety of MabThera SC (rituximab, subcutaneous) induction therapy in patients with non-Hodgkin's lymphoma, following a first initial treatment of MabThera IV (rituximab, intraveneous). Induction treatment period in the study is estimated to be 8 months.

ELIGIBILITY:
Inclusion Criteria:

1. Indication according to the Summary of Product Characteristics (SPC) for MabThera SC formulation:

   * As treatment of previously untreated patients with stage III-IV follicular lymphoma in combination with chemotherapy
   * As treatment of patients with CD20 positive diffuse large B cell non-Hodgkin's lymphoma in combination with chemotherapy
2. At least 4 treatment cycles with MabThera is planned
3. Patients >/= 18 years at inclusion
4. Patients written informed consent
5. Treatment decision to prescribe MabThera SC has been taken by the physician prior to recruitment into the study

Exclusion Criteria:

1. Contraindications according to SPC for MabThera SC formulation:

   * Hypersensitivity for the active substance or murine antibodies, hyaluronidase or any other excipients
   * Active and severe infections
   * Patients with severe immunsuppression
2. Patient included in clinical trials with experimental pharmaceuticals
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients within label indication for MabThera SC and subject for induction therapy with MabThera SC; patients object for maintenance therapy are excluded
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Response rate using the International Working Group criteria | 8 months

SECONDARY OUTCOMES:
Incidence of adverse events | Through to end of study, up to approximately 1 year
Incidence of administration related reactions during induction therapy in patients who have previously received at least one dose of MabThera IV | Through to end of study, up to approximately 1 year
Incidence of serious adverse events | Through to end of study, up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Sweden (7):
  - Eskilstuna
  - Halmstad
  - Helsingborg
  - Linköping
  - Luleå
  - Örebro
  - Visby